CLINICAL TRIAL: NCT01615445
Title: A Pilot Randomized Controlled Clinical Trial of Resveratrol Supplementation on Exercise in Healthy Sedentary Adults
Brief Title: Resveratrol Supplementation on Exercise in Healthy Sedentary Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2008540-01H
Record Dates: First submitted 2012-05-25; First posted 2012-06-08 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Active Comparator): Group A Participants will received resveratrol 500 mg twice daily for 1 week then 1000 mg twice daily for 3 weeks, according to tolerance. They will discontinue medication for 2 weeks. The will receive placebo for 4 weeks.
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Group B (n=6) Will receive placebo for 4 weeks, they will discontinue medication for two weeks. Then receive resveratrol for 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Resveratrol — Group A: resveratrol 1000 mg (500 mg twice) daily for 1 week then by tolerance and safety 2000 mg (1 000mg twice) daily for 3 weeks, followed by no medication for two weeks and then placebo for twice daily for 4 weeks.
  Arms: Resveratrol
Drug: placebo — Participants will receive placebo daily for 4 weeks, followed by no medication for two weeks and then resveratrol 1 000 mg(500 mg twice) daily for 1 week, then by tolerance and safety 2 000 mg (1 000 mg twice) daily for three weeks.
  Arms: Placebo

SUMMARY:
Previous animal studies have found that resveratrol supplementation significantly increased aerobic capacity. The investigators conducted a randomized placebo-controlled cross-over study to assess whether resveratrol could provide similar benefits in humans.

All participants were assigned to two 4-week treatment periods, with a 2 week washout in-between. During one period, volunteers in received resveratrol and during the other period, they received identical-appearing placebo.

The primary outcome of interest was change in exercise capacity, as measured by change in exercise duration on constant load exercise testing and change in aerobic capacity (peak VO2) on incremental exercise testing. Secondary outcomes were tolerability and side-effects associated with resveratrol.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 18-65 years
* healthy, sedentary as per CDC (Less than 150 minutes of moderate activity[brisk walking] or less than 75 minutes of strenuous activity [jogging] on a typical week)
* not planning a significant change in their level of physical activity during the study period
* have a body mass index (BMI) between 20 and 30
* give informed consent and be willing to comply with protocol requirements

Exclusion Criteria:

* have heart disease, lung disease, and liver disease
* be unable to perform maximal exercise on a cycle ergometer ("maximal" defined by attainment of peak heart rate or ventilation within 15% of the predicted maximum or a respiratory quotient of > 1.15). It should be noted that maximal does not imply normal aerobic capacity
* use medications that may affect exercise performance ( β-blockers, Ca channel blockers
* be a smoker or have a past history of smoking more than total 5 pkg/year
* be pregnant or lactating
* use oral contraceptives
* have severe or unstable medical illness
* have blood/urine screening test results outside of the normal reference range and deemed clinically significant by the clinical investigator. Note: only minor variations in screening results outside of the normal references ranges will be permitted.
* take an anticoagulant, antiplatelet, NSAID, antidiabetic, antihypertensive, estrogen, SERM, immunosuppressant, vasodilator drug; or a significant medication metabolized via cytochrome P450 enzymes
* have current or history of a hormonal disorder, including cancer
* have a bleeding disorder, autoimmune condition
* have allergies to any of the ingredients in the study product or placebo
* have thrombosis of lower extremities
* have electrolyte abnormalities
* have recent myocardial infarction (i.e. within one year or less)
* have unstable angina
* have uncontrolled arrhythmia's causing symptoms or haemodynamic compromise
* have active endocarditis
* have acute myocarditis or pericarditis
* have symptomatic severe aortic stenosis
* have uncontrolled heart failure
* have acute non-cardiac disorder that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis)
* have a left main coronary stenosis or its equivalent
* have moderate stenotic valvular heart disease
* have severe untreated arterial hypertension (>200 mmHg systolic, >120 mmHg diastolic)
* have significant pulmonary hypertension
* have tachyarrhythmias or bradyarrhythmias
* have hypertrophic cardiomyopathy
* have mental impairment leading to inability to cooperate
* have high-degree atrioventricular block
* have cardiac (bradyarrhythmias, ventricular tachycardia, myocardial infarction, heart failure, hypotension, and shock) and non-cardiac (musculoskeletal trauma, severe fatigue, dizziness, fainting, body aches) complications.
* have kidney disease
* have excessive vomiting
* be dehydrated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in duration of constant load exercise | Phase I: Baseline and 4 weeks; Phase II (cross-over phase): 6 weeks and 10 weeks
  The primary outcome would be the change in constant load exercise duration between baseline and follow-up visits, expressed as a percent change from the baseline constant load test. The average change from baseline will be compared between the experimental and control groups.
Change from baseline in aerobic capacity(peak VO2) | Phase I: Baseline and 4 weeks; Phase II (cross-over phase): 6 weeks and 10 weeks
  The aerobic capacity (peak VO2)is assessed by incremental exercise tests.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nha Voduc, MD, Principal Investigator — The Ottawa Hospital, The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital -General Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Voduc N, la Porte C, Tessier C, Mallick R, Cameron DW. Effect of resveratrol on exercise capacity: a randomized placebo-controlled crossover pilot study. Appl Physiol Nutr Metab. 2014 Oct;39(10):1183-7. doi: 10.1139/apnm-2013-0547. Epub 2014 Apr 30. PMID 25051174
- See also: click here to view trial results — http://www.nrcresearchpress.com/doi/abs/10.1139/apnm-2013-0547